CLINICAL TRIAL: NCT06239675
Title: Concurrent Transcranial Direct Current Stimulation and Constraint-induced Movement Therapy in Children With Hemiplegic Cerebral Palsy: A Randomized Controlled Study on Efficacy and Brain Mechanisms
Brief Title: Cerebral pAlsy Motor Promotion With Transcranial Direct Current Stimulation (CAMP-tDCS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funds are available to support implementation of this project.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Health (Other)
Responsible Party: Principal Investigator, Yanlong Song, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2023-0925
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy, Hemiplegic
Keywords: children
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Direct Current Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tDCS+CIMT (Experimental): Participants will receive concurrent anodal tDCS (20 minutes, 1mA~2mA) and CIMT (2 hours) five days a week for three weeks in a row.
  Interventions: Device: tDCS; Behavioral: CIMT
- sham+CIMT (Sham Comparator): Participants will receive concurrent sham tDCS and CIMT (2 hours) five days a week for three weeks in a row.
  Interventions: Behavioral: CIMT; Device: sham tDCS

INTERVENTIONS:
Device: tDCS — tDCS will be delivered anodal for 20 minutes at an intensity between 1mA and 2mA for 15 sessions.
  Other Names: transcranial direct current stimulation
  Arms: tDCS+CIMT
Behavioral: CIMT — CIMT will be administered for two hours a day, five days a week, and three weeks in a row.
  Other Names: constraint induced movement therapy
Device: sham tDCS — sham tDCS
  Arms: sham+CIMT

SUMMARY:
This study aims to test if transcranial direct current stimulation (tDCS) can be applied to boost the efficacy of constraint-induced movement therapy (CIMT) in children with HCP and examine brain mechanisms related to individual outcomes.

DETAILED DESCRIPTION:
Currently, clinical treatment of hand/arm motor deficits in children affected by cerebral palsy is mainly rehabilitation and behaviorally oriented. Constraint-induced movement therapy (CIMT) has emerged as a frequently used rehabilitation intervention in children with hemiplegic cerebral palsy (HCP). In CIMT sessions, the unaffected upper limb is restrained with a cast or similar device, and the affected hand/arm is intensively and structurally trained. With different variations, such as constraint and intensity, CIMT has been demonstrated to be efficacious in improving hand-and-arm use in children with HCP. However, clinical outcomes across individuals who receive CIMT can show vast variation. How to improve the efficacy of CIMT and reduce individual variation will be of direct and profound clinical impacts. Motor deficits of children with HCP have a source origin of early brain injury, which often disrupts some regions of the brain and can cause changes in brain functions. Alteration or normalization of brain neuronal activities may influence motor functions in children with HCP and might boost the efficacy of CIMT. Transcranial direct current stimulation (tDCS), a type of non-invasive weak electric stimulation, has been demonstrated to be capable of influencing cognition and behaviors in abundant laboratory research tasks, hinting at potential clinical effects. Specific to the pediatric population with HCP, a few preliminary studies have tested the safety of tDCS when applied in children with HCP. This study will test how tDCS influences the efficacy of CIMT in children with HCP by comparing motor performances between two groups. The first group of children with HCP will receive anodal tDCS and CIMT while the second group of children with HCP will receive sham tDCS and CIMT during the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* formal diagnosis of hemiplegic cerebral palsy
* unilateral upper limb (arm and hand) motor and sensory impairments
* capable of understanding and following experimental instructions and procedures
* capable of performing study procedures without assistance
* 5-17 years of age, including 5-year-old and 17-year-old

Exclusion Criteria:

* brain surgery, peripheral nerve surgery, genetic disorders, other neurological disorders or injuries
* muscle toxin injection within six months before recruitment
* received constraint-induced movement therapy (CIMT) within one year before recruitment
* uncontrolled seizures within one year before recruitment
* orthopedic surgery in upper limb within one year before recruitment
* incapable of understanding and following experimental instructions and procedures
* non-removable metallic objects or infusion pumps in the body
* psychoactive or myorelaxant medication during study procedures
* less than five years of age and older than 17 years of age

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
gross manual dexterity | With the first day of the intervention defined as day 1, this measure will be assessed in one of the three days before day 1, on day 15 or day 16 or day 17, and on day 181 or day 182 or day 183.
  It will be measured by the box and block test to assess how many blocks one can move from one box to another in one minute.
fine manual dexterity | With the first day of the intervention defined as day 1, this measure will be assessed in one of the three days before day 1, on day 15 or day 16 or day 17, and on day 181 or day 182 or day 183.
  It will be measured by the nine-hole peg test to assess the time one needs to place nine pins into a reservior.

SECONDARY OUTCOMES:
quality of upper extremity skill | With the first day of the intervention defined as day 1, this measure will be assessed in one of the three days before day 1, on day 15 or day 16 or day 17, and on day 181 or day 182 or day 183.
  It will be subjectively assessed with the Quality of Upper Extremity Skill Test (QUEST) to measure functions and use of both upper limbs.
finger touch sensitivity | With the first day of the intervention defined as day 1, this measure will be assessed in one of the three days before day 1, on day 15 or day 16 or day 17, and on day 181 or day 182 or day 183.
  It will be measured with a two-point discriminator to assess the minimal displacement between two points of touch on fingertip one can perceive.

CONTACTS AND LOCATIONS:
Overall Officials: Yanlong Song, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Health Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants' identifiers and linkages between study IDs and participants' identifiers will not be shared to protect participants' privacy, rights, and confidentiality. All other individual participant data will be preserved and shared. All data to be shared will be de-identified prior to receipt by any data repository. The information needed to generate a global unique identifier for a repository will be kept for each participant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be shared at the end of the study.
Access Criteria: Access to the shared IPD and supporting information will not be controlled.